CLINICAL TRIAL: NCT01942759
Title: The Prognostic Value of FDG PET/CT and Diffusion-weighed Imaging on Detection of Primary Tumor and Axillary Metastasis for Breast Cancer: SUVMax Against to ADC
Brief Title: The Prognostic Value of FDG PET/CT and Diffusion-weighed Imaging on Breast Cancer
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Aynur Ozen, Aynur Ozen, Bagcilar Training and Research Hospital
Other Study IDs: BC-PET-MR-01
Record Dates: First submitted 2013-09-02; First posted 2013-09-16 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Positron-Emission Tomography; Diffusion Magnetic Resonance Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Histologic grade: According to the modified criteria of Bloom and Richardson grading system: grade 1, 2 and 3
- Axillary metastasis: Group A: axillary lymph node metastasis Group B: no axillary lymphatic metastasis
- Modified Nottingham prognostic index: NPI = pathological tumour size (cm) × 0.2 + lymph node stage (1, 2 or 3) + histological grade (1, 2 or 3)
  The cut-off points of the index were 3.4 and 5.4 to divide patients into the good (≤3.4), moderate (3.41-5.4) and poor (>5.4) prognostic groups
- Oestrogen receptor status: Negative Positive
- Progesterone receptor status: Negative Positive
- HER-2 neu status: Negative Positive

SUMMARY:
The purpose of this study is to determine findings of positron emission tomography and diffusion weighted magnetic resonance in primary lesion and axillary metastasis of breast cancer and compare of two imaging modality in these patients.

DETAILED DESCRIPTION:
We aimed that to correlate both primary lesion 18F-fluorodeoxyglucose (FDG) maximum standardized uptake value (SUVmax) and diffusion-weighted imaging (DWI) apparent diffusion coefficient (ADC) with clinicopathological prognostic factors and compare the prognostic value of these indexes in breast cancer in this study. The evaluated and compared parameters are SUVmax and ADC according to age, tumour size, lymph node metastasis, receptor status, histologic grade, modified Nottingham prognostic index.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of breast cancer for which surgical intervention is planned

Exclusion Criteria:

* patients received neoadjuvant chemotherapy
* before breast surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationships between both SUVmax and ADC and clinicopathological prognostic factors | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: AYNUR OZEN, MD, Study Chair — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)